CLINICAL TRIAL: NCT04890145
Title: The RW-Precision-Coupler Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020VIB010
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Hearing Loss
Keywords: Vibrant Soundbridge System; RW-Precision-Coupler
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mild to severe hearing loss (Experimental)
  Interventions: Device: RW-Precision-Coupler

INTERVENTIONS:
Device: RW-Precision-Coupler — Implantation of the RW-Precision-Coupler together with FMT-VORP 503

SUMMARY:
The RW-Precision-Coupler Clinical Investigation is prospective, non-randomized, open label, single subjects repeated measures, longitudinal monocentric trial. The primary aim of this pre-market clinical investigation is to evaluate the clinical performance and safety of VSB together with the VSB RWP-Coupler in the treatment of hearing loss. As secondary aims are to evaluate the clinical performance of VSB together with RWP-Coupler by measuring Sound Field audiometry (SF), to evaluate the safety of VSB together with RWP-Coupler by measuring bone conduction (BC) thresholds and collecting and assessing adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Geographically and physically able to return to the investigational site for scheduled evaluations and follow-up appointments

  * Fluent in the German language
  * Persons of 18 years of age or older
  * Signed and dated informed consent before the start of any study-specific procedure
  * The physician must fully assess the potential risks and benefits for the patient prior to the decision to implant the RW-Precision-Coupler. The physician must exercise medical judgment and consider the patient's complete hospital record (also called medical history)
  * No previous active middle ear implant surgery performed in the implanted ear
  * The following indication for VORP503:

    * For a patient with sensorineural hearing loss, pure-tone air conduction threshold levels at or within the levels listed below:
    * For a patient with conductive or mixed hearing loss, pure tone bone-conduction threshold levels at or within the levels listed below:
    * A patient shall present with an ear anatomy that can facilitate positioning of the FMT in contact with a suitable vibratory structure of the ear.
    * A patient with sensorineural hearing loss shall be a current user of an acoustic hearing aid and have used this aid for at least 4 hours (average) per day for at least 3 months prior to evaluation, or shall not be able to wear or benefit from conventional hearing aids for medical reasons.
    * A patient shall be psychologically and emotionally stable with realistic expectations of the benefits and limitations of the Soundbridge

Exclusion Criteria:

* Simultaneous participation in another clinical trial (on device or on drug) which would interfere with the results of the study

  * Pregnancy or lactation
  * Contraindication for RWP-Coupler Sizer:

    * if a patient is known to be intolerant of the materials used in the RWP-Coupler.
    * if a patient is known to be intolerant of the materials used in the RWP-Coupler Sizer.
    * in case of a fixed stapes footplate.
  * Contraindication for VORP503:

    * A patient is known to be intolerant of the materials used in the implant (medical grade silicone elastomer, medical grade epoxy and titanium).
    * A patient with retrocochlear, or central auditory disorders.
    * A patient with nonresponsive active ear infection and/or chronic fluid in or about the ear.
    * A patient whose hearing loss has demonstrated an improving and decreasing fluctuation over a two-year period of 15 dB in either direction.
    * A patient with any physical, psychological, or emotional disorder that would interfere with surgery or the ability to perform on test and rehabilitation procedures.
    * A patient with a skin or scalp condition that may preclude attachment of the audio processor with a magnet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Freiburger Monosyllable Test | 6 months post-operative
  Investigate the improvement of unaided pre-activation Word Recognition Scores (WRS) to 6 months post-operation aided WRS with RW-Precision-Coupler

CONTACTS AND LOCATIONS:
Overall Officials: Lenarz Thomas, Prof. h.c. Dr., Principal Investigator — Medizinische Hochschule Hannover Klinik und Poliklinik für Hals-Nasen-Ohren-Heilkunde
Locations (1):
- Medical School Hannover, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No